CLINICAL TRIAL: NCT01594489
Title: Effect of Aminophylline on Contrast Induced Acute Kidney Injury in Patients With Acute Myocardial Infarction Treated With Primary Angioplasty
Brief Title: Aminophylline and Contrast Induced Nephropathy in Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Mauro Maioli, Medical Doctor, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prato0704
Record Dates: First submitted 2012-05-06; First posted 2012-05-09 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Aminophylline

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminophylline (Experimental): Additional Aminophylline therapy to hydration (sodium bicarbonate) and N-acetilcysteine
  Interventions: Drug: Aminophylline
- Control group (Active Comparator): Control group treated with hydration (sodium bicarbonate) and N-acetilcysteine
  Interventions: Drug: Hydration plus N-acetylcisteine

INTERVENTIONS:
Drug: Aminophylline — * 200 mg of aminophylline administrated intravenously as a short infusion, started in emergency department, before primary angioplasty and contrast medium administration
  * Sodium bicarbonate (154 mEq/L in dextrose and H20) 3mL/kg for 1 hour before contrast medium, followed by an infusion of 1 mL/kg/h for 12 hours after procedure
  * N-acetilcysteine: intravenous bolus of 1200 mg before angioplasty and 1200 mg twice daily for the 48 hours after PCI
  Arms: Aminophylline
Drug: Hydration plus N-acetylcisteine — * Sodium bicarbonate (154 mEq/L in dextrose and H20) 3mL/kg for 1 hour before contrast medium, followed by an infusion of 1 mL/kg/h for 12 hours after procedure
  * N-acetilcysteine: intravenous bolus of 1200 mg before angioplasty and 1200 mg twice daily for the 48 hours after PCI
  Arms: Control group

SUMMARY:
The purpose of this study is to determine whether additional therapy with Aminophylline to hydration with sodium bicarbonate and administration of N-acetylcysteine is more effective to prevent contrast induced acute kidney injury in patients undergoing primary coronary intervention for acute ST elevation myocardial infarction.

DETAILED DESCRIPTION:
Due to the clinical relevance of contrast acute kidney injury a large number of prophylactic procedures have been investigated. N-acetylcysteine and hydration with sodium bicarbonate are proved to be protective against contrast acute kidney injury. The adenosine-mediated afferent arteriolar vasoconstriction is a possible pathomechanism of renal impairment by contrast agent. It has been observed that aminophylline/theophylline, competitive adenosine antagonists, improves oxygen delivery to ischemic tissue, diminishes oxidative damage to renal tissue and may also scavenge free radicals.

The purpose of this study was to investigated whether the additional therapy with adenosine antagonist aminophylline reduces the incidence of contrast renal damage in high risk patients who have acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with AMI candidates for primary PCI presenting within 12 h of symptom onset with ST-segment elevation of more than 1 mm in at least two contiguous leads of the electrocardiogram

Exclusion Criteria:

* contrast medium administration within the previous 10 days,
* end-stage renal failure requiring dialysis,
* refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Contrast-Induced Acute Kidney Injury | 3 days
  Contrast-Induced Acute Kidney Injury is defined as an increase in serum creatinine of >=25% or 0.5 mg/dL over the baseline value within 3 days after the administration of the contrast medium

SECONDARY OUTCOMES:
Adverse clinical events | 1 month
  Adverse clinical events within 1 month including in-hospital death and need for dialysis or hemofiltration

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Maioli, MD, Principal Investigator — Cardiology Unit, Misericordia e Dolce Hospital, Prato, Italy
Locations (1):
- Ospedale Misericordia e Dolce, Prato, Prato, Italy